CLINICAL TRIAL: NCT02954731
Title: Trans-diagnostic Group CBT vs. Standard Group CBT for Depression, Social Anxiety and Agoraphobia/Panic Disorder: A Pragmatic, Multicenter Non-inferiority Randomized Controlled Trial
Brief Title: Trans-diagnostic Group CBT vs. Standard Group CBT for Depression, Social Anxiety and Agoraphobia/Panic Disorder
Acronym: TRACT-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Psychiatric Research Unit, Region Zealand, Denmark (Other)
Collaborators: Aarhus University Hospital (Other); Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Sidse Arnfred, Associate Professor, Consultant, Psychiatric Research Unit, Region Zealand, Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SA005
Record Dates: First submitted 2016-10-25; First posted 2016-11-03 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Depression, Unipolar; Anxiety Disorder Social; Panic Disorder
Keywords: Cognitive Behavior Therapy; Negative Affect; Unified Protocol; Session Tracking; Mechanisms of Change in Psychotherapy
MeSH Terms: conditions — Depressive Disorder; Phobia, Social; Panic Disorder

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- UP-CBT (Experimental): The "Unified Protocol for Transdiagnostic Treatment of Emotional Disorders" (UP) is one of the most widely studied transdiagnostic manuals. Here, the investigators apply a group manual that has been modified from the published UP for individual therapy based on recommendations on group delivery from the UP Institute (personal communications) and integrations modifications necessary for the delivery in the Mental Health Service. Group UP-CBT, consist of 8 treatment modules delivered in 14 group sessions given weekly in 2 hour sessions.
  Interventions: Behavioral: UP-CBT
- Standard-CBT (Active Comparator): Group CBT following Danish versions of diagnosis specific manuals (Social Anxiety Disorder (SAD) Group; Depression (DEP) Group; Agoraphobia/Panic Disorder (Ag/PD) (standard-CBT). The original elements of psychoeducation, cognitive restructuring, and exposure/activity scheduling are present in the applied manuals. Standard-CBT, consist of 8 treatment modules delivered in 14 group sessions given weekly in 2 hour sessions.
  Interventions: Behavioral: Standard-CBT

INTERVENTIONS:
Behavioral: UP-CBT — Psychotherapy in groups based on the "Unified Protocol" a third generation CBT-type psychotherapy
  Arms: UP-CBT
Behavioral: Standard-CBT — Psychotherapy in groups based on diagnosis specific, manualized, cognitive behavior therapy
  Arms: Standard-CBT

SUMMARY:
Transdiagnostic Cognitive Behavior Therapy (CBT) delivered in the individual format, have been proven just as effective as traditional diagnosis specific CBT manuals. The investigators have translated and modified the "The Unified Protocol for Transdiagnostic Treatment of Emotional Disorders" (UP-CBT) to make it applicable as group therapy in Danish Mental Health Service and a naturalistic trial of this manual has shown promising results. As the use of one manual instead of several diagnosis specific manuals in regional clinics could simplify logistics and reduce waiting time, the investigators want to compare group UP-CBT with diagnosis specific group CBT.

Method: A partial blinded, pragmatic, non-inferiority, multicentre randomized clinical trial (RCT). UP-CBT is compared to treatment-as-usual CT. 124 patients are included in each intervention arm, recruited from three Danish regional Mental Health Service Clinics. 31st July 2018 suppl: Inclusion number expanded to 170 in each arm due to unexpected large drop-out.

DETAILED DESCRIPTION:
Background: Transdiagnostic Cognitive Behavior Therapy (TCBT) Manuals delivered in individual format, have been reported to be just as effective as traditional diagnosis specific CBT manuals. The investigators have translated and modified the "The Unified Protocol for Transdiagnostic Treatment of Emotional Disorders" (UP-CBT) developed by Barlow and colleagues for use in Mental Health Service (MHS), and shown effects comparable to traditional CBT in a naturalistic trial. As the use of one manual instead of several diagnosis-specific manuals could simplify logistics, reduce waiting time, and increase therapist expertise compared to diagnosis specific CBT, the study aim to test the relative efficacy of group UP-CBT and diagnosis specific group CBT.

Methods/design: It is a partially blinded, pragmatic, non-inferiority, parallel, multi-center randomized controlled trial (RCT) of UP-CBT vs diagnosis specific CBT for depression, social anxiety disorder and agoraphobia/panic disorder. In both arms, the intervention consists of weekly group session for 14 weeks. In total, 248 patients are recruited from three regional MHS centers across the country and included in two intervention arms.31st July 2018 suppl: Inclusion number expanded to 340 due to unexpected large drop-out.

Outcomes are measured at end of therapy and at 6 months follow-up. Weekly patient-rated outcomes and group evaluations are collected for every session. Outcome assessors, blind to delivered intervention, will perform the observer-based symptom ratings, and fidelity assessors will monitor manual adherence.

Discussion: The current study will be the first RCT investigating the dissemination of the UP in a MHS setting and UP delivered in groups and including patients with depression. Hence the results are expected to add substantially to the evidence base for rational group psychotherapy in MHS. The planned moderator and mediator analyses could spur new hypotheses about mechanisms of change in psychotherapy and the association between patient characteristics and treatment effect.

ELIGIBILITY:
Inclusion Criteria:

Referred to Danish Mental Health Service

1. a principal DSM-5 diagnosis of Unipolar Depression (single episode or recurrent)(app. 50%), Social Anxiety Disorder (app. 25%), and Agoraphobia/Panic Disorder (app 25%)
2. the patient is currently not using any antidepressants or use accepted antidepressants (according to predefined list), which have been unchanged for at least 4 weeks before inclusion and no change in antidepressants is anticipated,
3. sufficient knowledge of the Danish language.

Exclusion Criteria:

1. risk of suicide is high according to clinicians or assessment researchers
2. alcohol or drug dependence,
3. cluster A or B (DSM-5) personality disorder diagnosed by intake clinicians or assessment researcher,
4. co-morbidity of pervasive developmental disorder, psychotic disorders, eating disorders, bipolar disorder, or severe physical illness,
5. psychopharmacological treatment other than those predefined as acceptable,
6. patient does not accept to stop the use of anxiolytics within the first four weeks of intervention.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 292 (Actual)
Dates: Start 2016-12; Primary Completion 2019-04-11 (Actual); Study Completion 2019-12-11 (Actual)

PRIMARY OUTCOMES:
WHO Well-Being Index (WHO-5) | Week 19 after allocation
  Self-rating questionnaire, 5 items on positive quality of life, web-based

SECONDARY OUTCOMES:
Hopkins Symptom Check List (SCL-25) | Week 19 after allocation
  Validated questionnaire - web-based
Work and Social Adjustment Scale (WSAS) | Week 19 after allocation
  Validated questionnaire - web-based
Hamilton Depression Rating Scale (HDRS) | Week 19 after allocation
  6-item HDRS based on telephone interview
Hamilton Anxiety Rating Scale (HARS) | Week 19 after allocation
  6-item HARS based on telephone interview

OTHER OUTCOMES:
Overall Anxiety Severity and Impairment Scale (OASIS) | Weekly, weeks 4-19 after allocation, before session
  Validated questionnaire
Overall Depression Severity and Impairment Scale (ODSIS) | Weekly, weeks 4-19 after allocation, before session
  Validated questionnaire
WHO Well-Being Index (WHO-5) | Weekly, weeks 4-19 after allocation, before session
  Validated questionnaire
Positive Affect and Negative Affect Schedule (PANAS) | Week 19 after allocation
  Validated questionnaire - web-based
Positive Affect and Negative Affect Schedule (PANAS) | Week 42-43 after allocation
  Validated questionnaire - web-based
Hopkins Symptom Check List (SCL-25) | Week 42-43 after allocation
  Validated questionnaire - web-based
Emotion Regulation Questionnaire (ERQ) | Week 19 after allocation
  Validated questionnaire - web-based
Emotion Regulation Questionnaire (ERQ) | Week 42-43 after allocation
  Validated questionnaire - web-based
WHO Well-Being Index (WHO-5) | Week 42-43 after allocation
  Self-rating questionnaire, 5 items on positive quality of life, web-based
Emotion Regulation Strategies Questionnaire (ERSQ) | Week 19 after allocation
  Validated questionnaire - web-based
Emotion Regulation Strategies Questionnaire (ERSQ) | Week 42-43 after allocation
  Validated questionnaire - web-based
Perseverative Thinking Questionnaire (PTQ) | Week 19 after allocation
  Validated questionnaire - web-based
Perseverative Thinking Questionnaire (PTQ) | Week 42-43 after allocation
  Validated questionnaires - web-based
Becks Depression inventory (BDI-II) | Week 19 after allocation
  Validated questionnaire - web-based
Becks Depression inventory (BDI-II) | Week 42-43 after allocation
  Validated questionnaire - web-based
Work and Social Adjustment Scale (WSAS) | Week 42-43 after allocation
  Validated questionnaire - web-based
Personality Inventory for DSM-5 - Short Form (PID-5 SF) Negative Affectivity and Detachment domain scores | Week 19 after allocation
  Validated questionnaire - web-based
Personality Inventory for DSM-5 - Short Form (PID-5 SF) Negative Affectivity and Detachment domain scores | Week 42-43 after allocation
  Validated questionnaire - web-based
Liebowitch Social Anxiety Scale (LSAS) | Week 19 after allocation
  Validated questionnaire - web-based
Liebowitch Social Anxiety Scale (LSAS) | Week 42-43 after allocation
  Validated questionnaire - web-based
Panic Disorder Severity Scale (PDSS) | Week19 after allocation
  Validated questionnaire - web-based
Panic Disorder Severity Scale (PDSS) | Week 42-43 after allocation
  Validated questionnaire - web-based
Mobility Inventory for Agoraphobia (MIA) | Week 19 after allocation
  Validated questionnaire - web-based
Mobility Inventory for Agoraphobia (MIA) | Week 42-43 after allocation
  Validated questionnaire - web-based
Hamilton Depression Rating Scale | Week 42-43 after allocation
  6-item HDRS based on telephone interview
Hamilton Anxiety Rating Scale | Week 42-43 after allocation
  6-item HARS based on telephone interview
Client Satisfaction Questionnaire | Week 43
  8-item validated questionnaire, web-based
Patient Evaluation of Group Therapy | Week 19
  Purpose-made questionnaire
Group Questionnaire - brief | Weekly, weeks 4-19 after allocation, after session
  8 items from validated questionnaire about group atmosphere
Therapist Ratings of session methods and atmosphere | Weekly, weeks 4-19 after allocation, after session
  Purpose-made questionnaire
Homework and Event Tracker | Weekly, weeks 4-19 after allocation, before session
  Purpose-made question for patients about homework and events previous week

CONTACTS AND LOCATIONS:
Overall Officials: Sidse MH Arnfred, MD,PhD,DMSc, Principal Investigator — Universityhospital Copenhagen, Psychiatry West, Mental Health Services Region Zealand
Locations (4):
- Denmark (4):
  - Psychotherapeutic Unit, Mental Health Centre Copenhagen, Copenhagen, Capital Region
  - Outpatient Clinic for Anxiety and Personality Disorders, Risskov, Central Region
  - Outpatient Clinic for Mania and Depression, Risskov, Central Region
  - Psychiatric Outpatient Clinic, Slagelse, Region Sjælland

IPD SHARING:
Plan to Share IPD: No
The datasets generated by the planned study will not be publicly available due to the rules of the Danish Data Protection Agency, but will be available from the corresponding author, after publication, on reasonable request and following signed confidentiality agreement with PI and the Danish Data Protection Agency Region Zealand.

REFERENCES:
- [Background] Reinholt N, Aharoni R, Winding C, Rosenberg N, Rosenbaum B, Arnfred S. Transdiagnostic group CBT for anxiety disorders: the unified protocol in mental health services. Cogn Behav Ther. 2017 Jan;46(1):29-43. doi: 10.1080/16506073.2016.1227360. Epub 2016 Oct 5. PMID 27705086
- [Background] Reinholt N, Krogh J. Efficacy of transdiagnostic cognitive behaviour therapy for anxiety disorders: a systematic review and meta-analysis of published outcome studies. Cogn Behav Ther. 2014;43(3):171-84. doi: 10.1080/16506073.2014.897367. Epub 2014 Mar 19. PMID 24646219
- [Background] Farchione TJ, Fairholme CP, Ellard KK, Boisseau CL, Thompson-Hollands J, Carl JR, Gallagher MW, Barlow DH. Unified protocol for transdiagnostic treatment of emotional disorders: a randomized controlled trial. Behav Ther. 2012 Sep;43(3):666-78. doi: 10.1016/j.beth.2012.01.001. Epub 2012 Jan 18. PMID 22697453
- [Background] Wilamowska ZA, Thompson-Hollands J, Fairholme CP, Ellard KK, Farchione TJ, Barlow DH. Conceptual background, development, and preliminary data from the unified protocol for transdiagnostic treatment of emotional disorders. Depress Anxiety. 2010 Oct;27(10):882-90. doi: 10.1002/da.20735. PMID 20886609
- [Derived] Niemeijer M, Reinholt N, Poulsen S, Bach B, Christensen AB, Eskildsen A, Hvenegaard M, Arendt M, Arnfred S. Trait and symptom change in group cognitive behaviour therapy for anxiety and depression. Clin Psychol Psychother. 2023 Sep-Oct;30(5):1058-1070. doi: 10.1002/cpp.2857. Epub 2023 Apr 27. PMID 37106559
- [Derived] Arnfred SM, Aharoni R, Hvenegaard M, Poulsen S, Bach B, Arendt M, Rosenberg NK, Reinholt N. Transdiagnostic group CBT vs. standard group CBT for depression, social anxiety disorder and agoraphobia/panic disorder: Study protocol for a pragmatic, multicenter non-inferiority randomized controlled trial. BMC Psychiatry. 2017 Jan 23;17(1):37. doi: 10.1186/s12888-016-1175-0. PMID 28114915

DOCUMENTS (2):
  • Study Protocol (2016-12-19): https://cdn.clinicaltrials.gov/large-docs/31/NCT02954731/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/31/NCT02954731/SAP_002.pdf